CLINICAL TRIAL: NCT03895203
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Active Reference (Adalimumab) Study Evaluating the Efficacy and Safety of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Test the Efficacy and Safety of Bimekizumab in the Treatment of Subjects With Active Psoriatic Arthritis
Acronym: BE OPTIMAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PA0010; 2017-002322-20 (EudraCT Number)
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bimekzumab dosage regimen (Experimental): Subjects randomized to this arm will receive assigned bimekizumab dosage regimen and placebo to maintain the blinding with adalimumab and placebo arms during the Treatment Period.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Adalimumab dosage regimen (Active Comparator): Subjects randomized to this arm will receive the assigned adalimumab dosage regimen during the Treatment Period.
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Double-Blind Treatment Period and will be reallocated to receive bimekizumab dosage regimen during the Maintenance Period.
  Interventions: Drug: Bimekizumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: BKZ; UCB4940
  Arms: Bimekzumab dosage regimen; Placebo
Drug: Adalimumab — Adalimumab will be administered according to the labeling recommendations.
  Other Names: HUMIRA®
  Arms: Adalimumab dosage regimen
Other: Placebo — Subjects will receive placebo at pre-specified time-points.
  Other Names: PBO
  Arms: Bimekzumab dosage regimen; Placebo

SUMMARY:
This is a study to demonstrate the clinical efficacy, safety and tolerability of bimekizumab administered subcutaneously (sc) compared with placebo in the treatment of subjects with active Psoriatic Arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the subject
* Subject is male or female at least 18 years of age
* Female subject must be postmenopausal, permanently sterilized or willing to use a highly effective method of contraception
* Documented diagnosis of adult-onset Psoriatic Arthritis (PsA) meeting the Classification Criteria for Psoriatic Arthritis (CASPAR) for at least 6 months prior to Screening with active PsA and must have at Baseline tender joint count (TJC) >=3 out of 68 and swollen joint count (SJC) >=3 out of 66
* Subject must be negative for rheumatoid factor and anti-cyclic citrullinated peptide (CCP) antibodies
* Subject must have at least 1 active psoriatic lesion(s) and/or a documented history of psoriasis (PSO)
* Subject must be a suitable candidate for treatment with adalimumab and has no contraindications to receive adalimumab as per the local label as assessed by the Investigator
* Subjects currently taking NSAIDs, cyclooxygenase 2 (COX-2) inhibitors, analgesics (including mild opioids), corticosteroids, methotrexate (MTX), leflunomide (LEF), sulfasalazine (SSZ), hydroxychloroquine (HCQ) AND/OR apremilast can be allowed if they fulfill specific requirements prior to study entry

Exclusion Criteria:

* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study
* Subjects with current or prior exposure to any biologics for the treatment of Psoriatic Arthritis (PsA) or Psoriasis (PSO)
* Subject has an active infection or a history of recent serious infections
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has a diagnosis of inflammatory conditions other than PSO or PsA. Subjects with a diagnosis of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease (IBD) are allowed as long as they have no active symptomatic disease at Screening or Baseline
* Subject had acute anterior uveitis within 6 weeks of Baseline
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer
* Subject has a form of PSO other than chronic plaque-type (eg, pustular, erythrodermic and guttate PSO, or drug-induced PSO)
* Presence of active suicidal ideation, or moderately severe major depression or severe major depression
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (136):
- United States (25):
  - Pa0010 50017, Phoenix, Arizona
  - Pa0010 50035, San Diego, California
  - Pa0010 50004, Tustin, California
  - Pa0010 50033, Palm Harbor, Florida
  - Pa0010 50037, Tampa, Florida
  - Pa0010 50039, Atlanta, Georgia
  - Pa0010 50028, Lexington, Kentucky
  - Pa0010 50015, Hagerstown, Maryland
  - Pa0010 50016, St Louis, Missouri
  - Pa0010 50029, Albuquerque, New Mexico
  - Pa0010 50010, Brooklyn, New York
  - Pa0010 50125, Charlotte, North Carolina
  - Pa0010 50040, Dayton, Ohio
  - Pa0010 50020, Duncansville, Pennsylvania
  - Pa0010 50006, Wyomissing, Pennsylvania
  - Pa0010 50008, Johnston, Rhode Island
  - Pa0010 50007, Orangeburg, South Carolina
  - Pa0010 50001, Jackson, Tennessee
  - Pa0010 50012, Memphis, Tennessee
  - Pa0010 50002, Austin, Texas
  - Pa0010 50049, Corpus Christi, Texas
  - Pa0010 50051, Houston, Texas
  - Pa0010 50036, Mesquite, Texas
  - Pa0010 50009, Waco, Texas
  - Pa0010 50050, Beckley, West Virginia
- Australia (6):
  - Pa0010 30005, Camberwell
  - Pa0010 30002, Clayton
  - Pa0010 30008, Hobart
  - Pa0010 30003, Maroochydore
  - Pa0010 30007, Victoria Park
  - Pa0010 30006, Woodville
- Belgium (3):
  - Pa0010 40003, Genk
  - Pa0010 40002, Leuven
  - Pa0010 40059, Mons
- Canada (4):
  - Pa0010 50041, Québec
  - Pa0010 50042, Rimouski
  - Pa0010 50043, Sidney
  - Pa0010 50044, Trois-Rivières
- Czechia (11):
  - Pa0010 40061, Brno
  - Pa0010 40065, Brno
  - Pa0010 40062, Ostrava
  - Pa0010 40009, Pardubice
  - Pa0010 40013, Prague
  - Pa0010 40014, Prague
  - Pa0010 40015, Prague
  - Pa0010 40063, Prague
  - Pa0010 40066, Prague
  - Pa0010 40010, Uherské Hradiště
  - Pa0010 40012, Zlín
- France (2):
  - Pa0010 40019, Paris
  - Pa0010 40068, Tours
- Germany (12):
  - Pa0010 40074, Bad Doberan
  - Pa0010 40025, Berlin
  - Pa0010 40028, Berlin
  - Pa0010 40076, Cottbus
  - Pa0010 40023, Erlangen
  - Pa0010 40117, Frankfurt
  - Pa0010 40029, Hamburg
  - Pa0010 40071, Hamburg
  - Pa0010 40027, Herne
  - Pa0010 40078, Leipzig
  - Pa0010 40348, Magdeburg
  - Pa0010 40026, Ratingen
- Hungary (8):
  - Pa0010 40081, Budapest
  - Pa0010 40083, Budapest
  - Pa0010 40032, Debrecen
  - Pa0010 40030, Eger
  - Pa0010 40082, Kistarcsa
  - Pa0010 40079, Szentes
  - Pa0010 40033, Székesfehérvár
  - Pa0010 40080, Szombathely
- Italy (4):
  - Pa0010 40084, Catania
  - Pa0010 40087, Milan
  - Pa0010 40085, Pisa
  - Pa0010 40086, Reggio Emilia
- Japan (14):
  - Pa0010 20035, Bunkyō City
  - Pa0010 20036, Kawachi-Nagano-shi
  - Pa0010 20045, Kita-ku
  - Pa0010 20049, Kitakyushu
  - Pa0010 20044, Minatoku
  - Pa0010 20033, Nagoya
  - Pa0010 20041, Osaka
  - Pa0010 20046, Osaka
  - Pa0010 20048, Saitama
  - Pa0010 20031, Sapporo
  - Pa0010 20042, Sasebo
  - Pa0010 20032, Suita
  - Pa0010 20043, tabashi City
  - Pa0010 20030, Tokyo
- Poland (19):
  - Pa0010 40093, Bialystok
  - Pa0010 40119, Bydgoszcz
  - Pa0010 40038, Elblag
  - Pa0010 40088, Elblag
  - Pa0010 40096, Gdynia
  - Pa0010 40042, Krakow
  - Pa0010 40092, Krakow
  - Pa0010 40037, Lublin
  - Pa0010 40091, Nowa Sól
  - Pa0010 40044, Poznan
  - Pa0010 40090, Poznan
  - Pa0010 40118, Torun
  - Pa0010 40041, Warsaw
  - Pa0010 40094, Warsaw
  - Pa0010 40097, Warsaw
  - Pa0010 40098, Warsaw
  - Pa0010 40039, Wroclaw
  - Pa0010 40043, Wroclaw
  - Pa0010 40095, Wroclaw
- Russia (17):
  - Pa0010 20002, Moscow
  - Pa0010 20005, Moscow
  - Pa0010 20010, Moscow
  - Pa0010 20017, Moscow
  - Pa0010 20013, Petrozavodsk
  - Pa0010 20012, Ryazan
  - Pa0010 20016, Ryazan
  - Pa0010 20001, Saint Petersburg
  - Pa0010 20003, Saint Petersburg
  - Pa0010 20004, Saint Petersburg
  - Pa0010 20009, Saint Petersburg
  - Pa0010 20083, Saint Petersburg
  - Pa0010 20007, Saratov
  - Pa0010 20014, Ulyanovsk
  - Pa0010 20006, Vladimir
  - Pa0010 20008, Yaroslavl
  - Pa0010 20015, Yaroslavl
- Spain (9):
  - Pa0010 40045, A Coruña
  - Pa0010 40105, Córdoba
  - Pa0010 40102, Málaga
  - Pa0010 40101, Sabadell
  - Pa0010 40104, Santiago de Compostela
  - Pa0010 40049, Seville
  - Pa0010 40103, Seville
  - Pa0010 40106, Seville
  - Pa0010 40099, Vigo
- United Kingdom (2):
  - Pa0010 40111, Leeds
  - Pa0010 40107, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Ritchlin CT, Coates LC, McInnes IB, Mease PJ, Merola JF, Tanaka Y, Asahina A, Gossec L, Gottlieb AB, Warren RB, Ink B, Bajracharya R, Shende V, Coarse J, Landewe RB. Bimekizumab treatment in biologic DMARD-naive patients with active psoriatic arthritis: 52-week efficacy and safety results from the phase III, randomised, placebo-controlled, active reference BE OPTIMAL study. Ann Rheum Dis. 2023 Nov;82(11):1404-1414. doi: 10.1136/ard-2023-224431. Epub 2023 Sep 11. PMID 37696588
- [Result] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Result] Kristensen LE, Tillett W, Nash P, Coates LC, Mease PJ, Ogdie A, Gisondi P, Ink B, Prickett AR, Bajracharya R, Taieb V, Lyris N, Lambert J, Walsh JA. Association of achieving clinical disease control criteria and patient-reported outcomes in bimekizumab-treated patients with active psoriatic arthritis: results from two phase III studies. Ther Adv Musculoskelet Dis. 2024 Nov 11;16:1759720X241288071. doi: 10.1177/1759720X241288071. eCollection 2024. PMID 39534481
- [Result] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Summary of Research: Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2025 Aug;12(4):609-612. doi: 10.1007/s40744-025-00764-8. Epub 2025 May 10. PMID 40347389
- [Result] Thaci D, Asahina A, Boehncke WH, Gottlieb AB, Lebwohl M, Warren RB, Edens H, Ink B, Bajracharya R, Coarse J, Merola JF. Bimekizumab Efficacy and Safety in Patients with Psoriatic Arthritis with Substantial Skin and Nail Psoriasis to 1 Year. Dermatol Ther (Heidelb). 2025 Dec 12. doi: 10.1007/s13555-025-01599-5. Online ahead of print. PMID 41381988
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Gladman DD, Mease PJ, Gossec L, Husni ME, Gottlieb AB, Ink B, Bajracharya R, Coarse J, Lyris N, Lambert J, Tillett W. Effect of Bimekizumab on Patient-Reported Outcomes and Work Productivity in Patients With Psoriatic Arthritis: 1-Year Results From 2 Phase III Studies. J Rheumatol. 2025 May 1;52(5):466-478. doi: 10.3899/jrheum.2024-0923. PMID 39892885
- [Derived] Husni ME, Mease PJ, Merola JF, Tillett W, Goldammer N, Ink B, Coarse J, Lambert J, Taieb V, Gladman DD. Bimekizumab provided rapid improvements in patient-reported symptoms and health-related quality of life in patients with active psoriatic arthritis: pooled 16-week results from two phase 3 studies. RMD Open. 2024 Sep 23;10(3):e004464. doi: 10.1136/rmdopen-2024-004464. PMID 39313302
- [Derived] Mease PJ, Merola JF, Tanaka Y, Gossec L, McInnes IB, Ritchlin CT, Landewe RBM, Asahina A, Ink B, Heinrichs A, Bajracharya R, Shende V, Coarse J, Coates LC. Safety and Efficacy of Bimekizumab in Patients with Psoriatic Arthritis: 2-Year Results from Two Phase 3 Studies. Rheumatol Ther. 2024 Oct;11(5):1363-1382. doi: 10.1007/s40744-024-00708-8. Epub 2024 Aug 31. PMID 39215949
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Risankizumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1403-1412. doi: 10.1007/s40744-024-00706-w. Epub 2024 Aug 9. PMID 39120849
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Ustekinumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Oct;11(5):1413-1423. doi: 10.1007/s40744-024-00705-x. Epub 2024 Aug 9. PMID 39120848
- [Derived] Gossec L, Orbai AM, de Wit M, Coates LC, Ogdie A, Ink B, Coarse J, Lambert J, Taieb V, Gladman DD. Effect of bimekizumab on patient-reported disease impact in patients with psoriatic arthritis: 1-year results from two phase 3 studies. Rheumatology (Oxford). 2024 Sep 1;63(9):2399-2410. doi: 10.1093/rheumatology/keae277. PMID 38754125
- [Derived] Warren RB, McInnes IB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, Mease PJ. Comparative Effectiveness of Bimekizumab and Guselkumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):829-839. doi: 10.1007/s40744-024-00659-0. Epub 2024 Mar 15. PMID 38488975
- [Derived] Maloney A, Dua P, Ahmed GF. Comparative Effectiveness of Bimekizumab in Psoriatic Arthritis: A Model-Based Meta-Analysis of American College of Rheumatology Response Criteria. Clin Pharmacol Ther. 2024 May;115(5):1007-1014. doi: 10.1002/cpt.3135. Epub 2024 Jan 12. PMID 38073049
- [Derived] McInnes IB, Asahina A, Coates LC, Landewe R, Merola JF, Ritchlin CT, Tanaka Y, Gossec L, Gottlieb AB, Warren RB, Ink B, Assudani D, Bajracharya R, Shende V, Coarse J, Mease PJ. Bimekizumab in patients with psoriatic arthritis, naive to biologic treatment: a randomised, double-blind, placebo-controlled, phase 3 trial (BE OPTIMAL). Lancet. 2023 Jan 7;401(10370):25-37. doi: 10.1016/S0140-6736(22)02302-9. Epub 2022 Dec 6. PMID 36493791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2019 and concluded in July 2022.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS) and Active Treatment-Blind Set (ATS).
Groups:
- Placebo: Participants received placebo during the 16-weeks Double-Blind Treatment Period (DBP).
- BKZ 160 mg Q4W: Participants received Bimekizumab (BKZ) 160 milligrams (mg) subcutaneous (SC) every 4 weeks (Q4W) during the 16-weeks DBP.
- ADA 40 mg Q2W: Participants received Adalimumab (ADA) 40 mg SC every 2 weeks (Q2W) during the 16-weeks DBP.
- Placebo/BKZ 160 mg Q4W: After the 16-weeks DBP, participants initially randomized to placebo received BKZ 160 mg SC Q4W during the 36-weeks Active Treatment-Blind Period (ATP).
- BKZ 160 mg Q4W/BKZ 160 mg Q4W: After the 16-weeks DBP, participants initially randomized to BKZ 160 mg continued to receive BKZ 160 mg SC Q4W during the 36-weeks ATP.
- ADA 40 mg Q2W/ADA 40 mg Q2W: After the 16-weeks DBP, participants initially randomized to ADA 40 mg continued to receive ADA 40 mg SC Q2W during the 36-weeks ATP.
Period: Double-Blind Treatment Period: 16 Weeks
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
Started | 281 | 431 | 140 | 0 | 0 | 0
Enthesitis at Baseline: PA0010/PA0011 Pooled Population | 106 | 249 | 0 | 0 | 0 | 0
Dactylitis at Baseline: PA0010/PA0011 Pooled Population | 47 | 90 | 0 | 0 | 0 | 0
Completed | 271 | 415 | 137 | 0 | 0 | 0
Not Completed | 10 | 16 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 8 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 1 | 0 | 0 | 0
Not completed — PHQ-9 Score elevated | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Site terminated | 0 | 1 | 0 | 0 | 0 | 0
Period: Active Treatment-Blind Period: 36 Weeks
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
Started | 0 | 0 | 0 | 271 | 414 (Eligible participants who continued to receive active treatment at Week 16 (participants not on treatment at Week 16 but continued in the study were excluded) were started in ATP.) | 136 (Eligible participants who continued to receive active treatment at Week 16 (participants not on treatment at Week 16 but continued in the study were excluded) were started in ATP.)
Completed | 0 | 0 | 0 | 257 | 387 | 125
Not Completed | 0 | 0 | 0 | 14 | 27 | 11
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 9 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 6 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 9 | 2
Not completed — COVID-19 Pandemic Circumstances | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal due to Subject Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Moving Out of Area | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the RS which consists of enrolled participants that have been randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Total
Number analyzed (Participants) | 281 | 431 | 140 | 852
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 255 | 386 | 122 | 763
  >=65 years | 26 | 45 | 18 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (11.7) | 48.5 (12.6) | 49.0 (12.8) | 48.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 230 | 69 | 453
  Male | 127 | 201 | 71 | 399
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 0 | 1 | 0 | 1
  Asian | 7 | 17 | 4 | 28
  Black | 0 | 1 | 1 | 2
  White | 270 | 410 | 133 | 813
  Other/mixed | 4 | 1 | 0 | 5
  Missing | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 2 | 11
  Not Hispanic or Latino | 276 | 426 | 136 | 838
  Missing | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Week 16
Description: ACR50 response rate: 50% or greater improvement of arthritis relative to Baseline. Those who met following 3 conditions for improvement from Baseline were classified as meeting ACR50 response criteria: greater than or equal (≥) 50% improvement in 68-tender joint count; ≥ 50% improvement in 66-swollen joint count; ≥ 50% improvement in at least 3 of 5 following parameters: Physician global assessment of disease activity (0-100 millimeter [mm] visual analog scale [VAS] [0 = no symptoms;100 = severe symptoms]), Patient global assessment of disease activity (100 mm VAS [0 = no limitation of normal activities; 100 = very poor]), Patient assessment of pain (100 mm VAS [0 = no pain; 100 = most severe pain]), Health Assessment Questionnaire-Disability Index (HAQ-DI) assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, lower scores indicated less disability and high-sensitivity C-reactive protein (hsCRP).
Time Frame: Week 16
Population: RS consisted of all enrolled participants who had been randomized. Participants who had missing ACR50 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not were considered as non-responders. Inferential Statistics for ADA 40 mg reference arm was not calculated and reported as no formal comparison was planned.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
percentage of participants | 10.0 | 43.9 | 45.7
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.082, 95% CI 2-sided [4.583 to 10.943]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 16 for Placebo and BKZ
Description: The HAQ-DI contains 20 items that measured the degree of difficulty experienced in the following 8 categories of the daily living activities: dressing and grooming (2 items), arising (2 items), eating (3 items), walking (2 items), hygiene (3 items), reach (2 items), grip (3 items), and common daily activities (3 items). Each question was scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). The overall HAQ-DI total score was calculated by dividing the sum of the highest category scores (0 to 24) by the number of categories with at least 1 question answered. The HAQ-DI total score ranges from 0 (no difficulty) to 3 (maximum difficulty). A lower HAQ-DI score indicated an improvement in function. Change from baseline was computed as the value at Week 16 minus the baseline value. A negative value in change from baseline indicated an improvement.
Time Frame: Baseline, Week 16
Population: RS consisted of all enrolled participants who had been randomized. Missing data and non-missing data preceded by a study treatment discontinuation were imputed using reference based multiple imputation. Descriptive statistics for ADA 40 mg reference arm was not calculated and reported since reference based imputation analysis method is used with Placebo as reference. As pre-specified in the SAP, this analysis was performed only for the participants randomized to Placebo and BKZ.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 281 | 431
score on a scale | -0.0881 (0.0273) | -0.2567 (0.0208)
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; Least square (LS) mean difference = -0.187, 95% CI 2-sided [-0.249 to -0.125]

3. Secondary Outcome: Percentage of Participants With a Psoriasis Area Severity Index (PASI) 90 Response at Week 4 in the Subgroup of Participants With Psoriasis (PSO) Involving at Least 3% Body Surface Area (BSA) at Baseline
Description: The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI = average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0 = no disease, the maximum score is 72 = maximal disease.
Time Frame: Baseline, Week 4
Population: Subset of study participants in RS with psoriasis involving at least 3% BSA at Baseline. Participants who have missing PASI90 data at Week 4 or who discontinued study treatment before Week 4 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 140 | 217 | 68
percentage of participants | 4.3 | 19.8 | 7.4

4. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 16 in the Subgroup of Participants With PSO Involving at Least 3% BSA at Baseline
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Subset of study participants in RS with psoriasis involving at least 3% BSA at Baseline. Participants who have missing PASI90 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they have data or not are considered as non-responders. Inferential Statistics for ADA 40 mg reference arm was not calculated and reported as no formal comparison was planned.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 140 | 217 | 68
percentage of participants | 2.9 | 61.3 | 41.2
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 63.039, 95% CI 2-sided [22.211 to 178.918]

5. Secondary Outcome: Change From Baseline in the Short Form 36-item Health Survey (SF-36) Physical Component Summary (PCS) at Week 16 for Placebo and BKZ
Description: SF-36 (version 2, standard recall):36-item generic health-related Quality of Life instrument that uses recall period of 4 weeks. Questionnaire has 36 questions composing scale that represent 8 domains:physical functioning; role physical; bodily pain;general health;vitality; social functioning;role emotional; and mental health. Scores for 8 domains were combined into two summary scores: physical component summary (PCS) score and mental component summary (MCS) score. Scores for 2 components summary (PCS and MCS) and 8 domains have been calculated and computed as raw/observed score to norm-based T-score metric(mean=50, standard deviation=10), raw score min=0(worst), max=100(best). Individual respondent's score falls outside T-score range of 45 to 55 was considered outside average range and when considering group-level data, score below 47 was considered indicative of impaired functioning within that health domain or dimension. Positive value in change from Baseline indicated improvement.
Time Frame: Baseline, Week 16
Population: RS consisted of all enrolled participants who had been randomized. Missing data and non-missing data preceded by a study treatment discontinuation were imputed using reference based multiple imputation. Descriptive statistics for ADA 40 mg reference arm was not calculated and reported since imputation analysis method was used with Placebo as reference. As pre-specified in the SAP, this analysis was performed only for the participants randomized to Placebo and BKZ.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 281 | 431
score on a scale | 2.326 (0.478) | 6.219 (0.402)
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS mean difference = 4.337, 95% CI 2-sided [3.229 to 5.444]

6. Secondary Outcome: Percentage of Participants With a Minimal Disease Activity (MDA) at Week 16
Description: MDA is measure to indicate disease remission, and is based on composite score of 7 domains. Participant is considered having achieved MDA if participant fulfills at least 5 of following 7 criteria: Tender joint count (0-68 joints) less than or equal to (≤1); Swollen joint count (0-66 joints) ≤ 1; PASI ≤ 1 or BSA ≤ 3: In PASI, body divided into four parts, head and neck, upper limb, trunk and lower limbs. Each area assessed for erythema, induration and scaling, each rated on a scale of 0 to 4. Total score ranges from 0(no disease) to 72 (maximal disease)]; Patient's Assessment of Arthritis Pain ≤ 15 [using VAS on a scale of 0 (no pain) to 100 (severe pain)]; Patient's Global Assessment of Disease Activity ≤ 20 [using VAS on a scale of 0 (very well) to 100 (very poor)]; HAQ-DI score ≤ 0.5, HAQ-DI score ranges from 0 (no difficulty) to 3 (maximum difficulty); Leeds Enthesitis Index score ≤ 1 for participants with enthesitis at baseline.
Time Frame: Week 16
Population: RS consisted of all enrolled participants who had been randomized. Participants who have missing MDA at Week 16 or who discontinued study treatment before Week 16 regardless of whether they have data or not are considered as non-responders. Inferential Statistics for ADA 40 mg reference arm was not calculated and reported as no formal comparison was planned.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
percentage of participants | 13.2 | 45.0 | 45.0
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.447, 95% CI 2-sided [3.668 to 8.088]

7. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (vdHmTSS) in Participants With Elevated Hs-CRP and/or at Least 1 Bone Erosion at Baseline at Week 16 for Placebo and BKZ
Description: The degree of joint damage was assessed using the vdHmTSS by quantifying the extent of bone erosions and joint space narrowing for 64 and 52 joints, respectively. The vdHmTSS ranges from 0 to 528, with higher scores representing greater damage. Descriptive statistics for ADA 40 mg reference arm was not calculated and reported since reference based imputation analysis method is used with Placebo as reference. As pre-specified in the SAP, this analysis was performed only for the participants randomized to Placebo and BKZ.
Time Frame: Baseline, Week 16
Population: Radiographic Set (RAS): all participants in RS who received at least 1 dose of investigational medicinal product (IMP) and have valid radiographic image of hands and feet (with assessment performed by at least 2 reviewers) at Screening. Missing data and non-missing data preceded by treatment discontinuation were imputed using reference based multiple imputation. Here, number of participants analyzed included RAS with elevated hs-CRP and/or with at least one bone erosion at Baseline.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 227 | 361
score on a scale | 0.36 (0.10) | 0.04 (0.05)
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p = 0.001, ANOVA; LS mean difference = -0.327, 95% CI 2-sided [-0.524 to -0.130]

8. Secondary Outcome: Percentage of Participants With an Enthesitis-free State in the Leeds Enthesitis Index (LEI) at Week 16 in the Subgroup of Participants With Enthesitis at Baseline in the Pooled Population of PA0010 and PA0011
Description: Presence of enthesitis was assessed in the subgroup of participants with enthesitis by palpation on the lateral epicondyles of the humerus (elbows), medial femoral epicondyles (knees), and Achilles tendons (heels) bilaterally and scored as 0 (no tenderness) and 1 (tenderness) at Baseline. The LEI consists of 6 items, 3 for the right part and 3 for the left part of the body. LEI is derived as the sum of the enthesitis score over the 6 sites mentioned above. The total score ranges from 0 to 6, higher scores indicates greater degree of enthesitis. Descriptive/Inferential statistics for ADA 40 mg reference arm was not calculated and reported since pooled data with PA0011 study is used which did not have ADA 40 mg arm.
Time Frame: Baseline of PA0010 for Participants of PA0010 and Baseline of PA0011 for Participants of PA0011, Week 16
Population: As pre-specified in the SAP, the subgroup of participants with enthesitis at Baseline in the pooled population of PA0010 and PA0011 (NCT03896581) were included for the analysis of outcome measure. Participants who have missing LEI at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as non achieving entheistis free-state.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 106 | 249
percentage of participants | 34.9 | 49.8
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 1.904, 95% CI 2-sided [1.180 to 3.074]

9. Secondary Outcome: Percentage of Participants With a Dactylitis-free State Based on the Leeds Dactylitis Index (LDI) at Week 16 in the Subgroup of Participants With Dactylitis at Baseline in the Pooled Population of PA0010 and PA0011
Description: The LDI quantitatively measures dactylitis using the circumference of involved digits and control digits and tenderness of involved digits. Digits affected by dactylitis are defined as those with a 10% difference in the ratio of circumference of the affected digit to the contralateral digit. The control digit is either the contralateral digit (digit on opposite hand or foot). The ratio of circumference between an affected digit and the control digit is multiplied by the tenderness score for the affected digit. The results from each involved digit are summed to provide the final LDI score. A higher LDI indicates worse dactylitis. Tenderness score (0 = no tenderness, 1 = tender). Descriptive/Inferential statistics for ADA 40 mg reference arm was not calculated and reported since pooled data with PA0011 study was used which did not have ADA 40 mg arm.
Time Frame: Baseline of PA0010 for Participants of PA0010 and Baseline of PA0011 for Participants of PA0011, Week 16
Population: As pre-specified in the SAP, the subgroup of participants with dactylitis at Baseline in the pooled population of PA0010 and PA0011 (NCT03896581) were included for the analysis of outcome measure. Participants who have missing LDI at Week 16 or who discontinued study treatment before Week 16 regardless of whether they have data or not are considered as non achieving dactylitis free-state.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 47 | 90
percentage of participants | 51.1 | 75.6
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.437, 95% CI 2-sided [1.559 to 7.574]

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Week 16
Description: The ACR20 response rate was based on a 20% or greater improvement of arthritis relative to Baseline. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria: 1. ≥ 20% improvement in 68-tender joint count; 2. ≥ 20% improvement in 66-swollen joint count; and 3. ≥ 20% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity (100 mm VAS [0 = no symptoms; 100 = severe symptoms]), Patient global assessment of disease activity (100 mm VAS [0 = no limitation of normal activities; 100 = very poor]), Patient assessment of pain (100 mm VAS [0 = no pain; 100 = most severe pain]), HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, lower scores indicated less disability, hsCRP.
Time Frame: Week 16
Population: RS consisted of all enrolled participants who had been randomized. Participants who have missing ACR20 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they have data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
percentage of participants | 23.8 | 62.2 | 68.6

11. Secondary Outcome: Change From Baseline in Van Der Heijde Modified Total Sharp Score (vdHmTSS) in the Overall Population at Week 16 for Placebo and BKZ
Description: The degree of joint damage was assessed using the vdHmTSS by quantifying the extent of bone erosions and joint space narrowing for 64 and 52 joints, respectively. The vdHmTSS ranges from 0 to 448, with higher scores representing greater damage. Descriptive statistics for ADA 40 mg reference arm was not calculated and reported since reference based imputation analysis method was used with Placebo as reference.
Time Frame: Baseline, Week 16
Population: The RAS consisted of all participants in the randomized set who received at least 1 dose of IMP and have a valid radiographic image of the hands and feet (with an assessment performed by at least the 2 reviewers) at Screening. Missing data and non-missing data preceded by a study treatment discontinuation were imputed using reference based multiple imputation. As pre-specified in the SAP, this analysis was performed only for the participants randomized to Placebo and BKZ.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W
Number analyzed (Participants) | 269 | 420
score on a scale | 0.32 (0.09) | 0.04 (0.04)
Statistical Analysis 1: Comparison: Placebo vs BKZ 160 mg Q4W; Test type: Superiority; p = 0.001, ANCOVA; LS mean difference = -0.281, 95% CI 2-sided [-0.452 to -0.111]

12. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 70 Response at Week 16
Description: The ACR70 response rate was based on a 70% or greater improvement of arthritis relative to Baseline. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria: 1. ≥ 70% improvement in 68-tender joint count; 2. ≥ 70% improvement in 66-swollen joint count; and 3. ≥ 70% improvement in at least 3 of the 5 following parameters: Physician global assessment of disease activity (100 mm VAS [0 = no symptoms;100 = severe symptoms]), Patient global assessment of disease activity (100 mm VAS [0 = no limitation of normal activities;100 = very poor]), Patient assessment of pain (100 mm VAS [0 = no pain; 100 = most severe pain]), HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), its score (0-3) computed from item scores, lower scores indicated less disability, hsCRP.
Time Frame: Week 16
Population: RS consisted of all enrolled participants who had been randomized. Participants who had missing ACR70 data at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
percentage of participants | 4.3 | 24.4 | 27.9

13. Secondary Outcome: Percentage of Participants With Investigator Global Assessment (IGA) Response Defined as Score of 0 (Clear) or 1 (Almost Clear) AND at Least a 2-grade Reduction From Baseline at Week 4 in the Subset of Participants With Psoriatic Skin Lesions at Baseline
Description: IGA measured the overall severity of PSO using the following 5-point scale and score was rated as 0 = clear (No signs of PSO; post-inflammatory hyperpigmentation may be present), 1 = almost clear (No thickening; normal to pink coloration; no to minimal focal scaling), 2 = mild (Just detectable to mild thickening; pink to light red coloration; predominately fine scaling), 3 = moderate (Clearly distinguishable to moderate thickening; dull to bright red, moderate scaling), and 4 = severe (Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions). The IGA response is defined as score of 0 (clear) or 1 (almost clear) with at least a 2-category improvement relative to Baseline.
Time Frame: Baseline, Week 4
Population: Subset of study participants in RS with psoriatic skin lesions at Baseline (minimal IGA score of 2) and with PSO involving at least 3% BSA at Baseline. Participants who had missing data at the Week 4 or who discontinued study treatment before or at the Week 4 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 129 | 204 | 62
percentage of participants | 3.9 | 28.9 | 11.3

14. Secondary Outcome: Percentage of Participants With an IGA Response Defined as Score of 0 (Clear) or 1 (Almost Clear) AND at Least a 2-grade Reduction From Baseline at Week 16 in the Subset of Participants With Psoriatic Skin Lesions at Baseline
Description: as for outcome 13
Time Frame: Baseline, Week 16
Population: Subset of study participants in RS with psoriatic skin lesions at Baseline (minimal IGA score of 2) and with PSO involving at least 3% BSA at Baseline. Participants who had missing data at the Week 16 or who discontinued study treatment before or at the Week 16 regardless of whether they had data or not are considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 129 | 204 | 62
percentage of participants | 3.9 | 50.5 | 33.9

15. Secondary Outcome: Change From Baseline in the Patient's Assessment of Arthritis Pain (PtAAP) at Week 16
Description: The PtAAP VAS is part of the American College of Rheumatology core set of measures in arthritis. Participants assessed their arthritis pain using a VAS ranging from 0 (no pain) to 100 (most severe pain). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: RS consisted of all enrolled participants who had been randomized. Missing data and non-missing data preceded by a study treatment discontinuation were imputed using reference based multiple imputation.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
score on a scale | -6.3 (1.5) | -23.6 (1.3) | -25.7 (2.5)

16. Secondary Outcome: Percentage of Participants With an Enthesitis-free State Based on the Spondyloarthritis Research Consortium of Canada (SPARCC) Index at Week 16 in the Subgroup of Participants With Enthesitis at Baseline
Description: Presence of enthesitis was assessed in the subgroup of participants with enthesitis at Baseline. The SPARCC index measures the severity of enthesitis through the assessment of 16 sites, 8 for the right part and 8 for the left part of the body: the greater trochanter (right/left), quadriceps tendon insertion into the patella (right/left), patellar ligament insertion into the patella and tibial tuberosity (right/left), achilles tendon insertion (right/left), plantar fascia insertion (right/left), medial and lateral epicondyles (right/left), and the supraspinatus insertion (right/left). Tenderness on examination is recorded as either present (1) or absent (0) for each of the 16 sites, for an average range of 0 (no enthesitis) to 16 (severe enthesitis).
Time Frame: Baseline, Week 16
Population: Subset of study participants in RS with SPARCC > 0 at Baseline. Participants who had missing SPARCC at Week 16 or who discontinued study treatment before Week 16 regardless of whether they had data or not are considered as not achieving enthesitis free-state.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 90 | 166 | 44
percentage of participants | 35.6 | 50.0 | 52.3

17. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease-12 (PsAID-12) Total Score at Week 16
Description: The PsAID-12 is a patient-reported outcome measure for assessing the impact of Psoriatic Arthritis (PsA) in 12 physical and psychological domains, including pain, fatigue, skin problems, work and/or leisure activities, functional capacity, discomfort, sleep disturbance, coping, anxiety/fear/uncertainty, embarrassment and/or shame, social participation, and depression. Each domain is assessed with a single question using a 0 to 10 numerical rating scale. Each domain score was multiplied by a weighting factor and the results were then summed to provide the total score. The total score ranged from 0 to 10, with higher scores indicating a worse status. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 15
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140
score on a scale | -0.53 (0.10) | -1.83 (0.09) | -2.14 (0.16)

18. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participants administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and within 140 days after the final dose of IMP.
Time Frame: From Baseline until Safety Follow-Up (up to Week 72)
Population: The Safety Set consisted of all participants who received at least 1 dose of the IMP. The ATS consisted of all participants who received at least 1 dose of active treatment (BKZ or ADA) during the ATP (Week 16 and after).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140 | 271 | 414 | 136
percentage of participants | 49.5 | 59.6 | 59.3 | 70.5 | 72.0 | 68.4

19. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: A SAE is any untoward medical occurrence that at any dose: Results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization; is a congenital anomaly or birth defect; is an infection that requires treatment parenteral antibiotics, other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and within 140 days after the final dose of IMP.
Time Frame: From Baseline until Safety Follow-Up (up to Week 72)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140 | 271 | 414 | 136
percentage of participants | 1.1 | 1.9 | 1.4 | 5.9 | 5.6 | 6.6

20. Secondary Outcome: Percentage of Participants With TEAEs Leading to Withdrawal From IMP During the Study
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participants administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and within 140 days after the final dose of IMP.
Time Frame: From Baseline until Safety Follow-Up (up to Week 72)
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
Number analyzed (Participants) | 281 | 431 | 140 | 271 | 414 | 136
percentage of participants | 1.1 | 1.9 | 2.1 | 1.8 | 2.7 | 3.7

ADVERSE EVENTS:
Time Frame: From Baseline until Safety Follow-Up (up to Week 72)
Description: TEAEs were defined as any AEs with an onset date on or after the date of first IMP administration and within 140 days after the final dose of IMP. TEAEs were analyzed and reported for Double-Blind Treatment Period (safety set) and Active Treatment-Blind Period (ATS) separately.
Arm/Group | Placebo | BKZ 160 mg Q4W | ADA 40 mg Q2W | Placebo/BKZ 160 mg Q4W | BKZ 160 mg Q4W/BKZ 160 mg Q4W | ADA 40 mg Q2W/ADA 40 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/431 | 0/140 | 1/271 | 0/414 | 0/136
Serious Adverse Events (participants affected / at risk) | 3/281 | 8/431 | 2/140 | 16/271 | 23/414 | 9/136
Other Adverse Events (participants affected / at risk) | 34/281 | 77/431 | 13/140 | 54/271 | 82/414 | 15/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=281) | BKZ 160 mg Q4W (N=431) | ADA 40 mg Q2W (N=140) | Placebo/BKZ 160 mg Q4W (N=271) | BKZ 160 mg Q4W/BKZ 160 mg Q4W (N=414) | ADA 40 mg Q2W/ADA 40 mg Q2W (N=136)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enchondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vascular disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Deep vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=281) | BKZ 160 mg Q4W (N=431) | ADA 40 mg Q2W (N=140) | Placebo/BKZ 160 mg Q4W (N=271) | BKZ 160 mg Q4W/BKZ 160 mg Q4W (N=414) | ADA 40 mg Q2W/ADA 40 mg Q2W (N=136)
Nasopharyngitis (Infections and infestations) | 13 (14) | 40 (44) | 7 (8) | 23 (28) | 29 (31) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 18 (18) | 22 (25) | 3 (3) | 12 (15) | 20 (21) | 5 (7)
Oral candidiasis (Infections and infestations) | 0 (0) | 9 (10) | 0 (0) | 14 (14) | 19 (26) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 9 (9) | 3 (3) | 15 (17) | 20 (20) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03895203/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT03895203/SAP_001.pdf